CLINICAL TRIAL: NCT01770834
Title: A Prospective, Non-interventional Multi-center Observational Study to Evaluate the Safety and Efficacy of Tocilizumab in Patients With Moderate to Severe Active Rheumatoid Arthritis in Routine Practice
Brief Title: A Prospective, Non-Interventional Study of RoActemra/Actemra (Tocilizumab) in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25533
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, observational study will evaluate the efficacy, safety and tolerability of RoActemra/Actemra (tocilizumab) in patients with moderate to severe active rheumatoid arthritis who have had an inadequate response or are intolerant to one or more conventional disease-modifying anti-rheumatic drugs. Data will be collected from patients initiated on RoActemra/Actemra treatment according to the local label at baseline, Weeks 4, 12 and 24, and at 3 and 6 months after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 21 years of age
* Moderate to severe active rheumatoid arthritis (DAS28 >/= 3.2)
* Inadequate response to one or more conventional disease-modifying anti-rheumatic drugs (DMARDs)
* Initiated on RoActemra/Actemra treatment in accordance with the prescribing information

Exclusion Criteria:

* Pregnant or lactating women
* Contra-indication to RoActemra/Actemra treatment according to the local labelling
* Previous treatment with tocilizumab
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* Women of childbearing potential not using effective methods of contraception as defined by protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe rheumatoid arthritis and an inadequate response or intolerant to previous therapy with conventional DMARDs
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04-18 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3 years

SECONDARY OUTCOMES:
Percentage of patients achieving a clinically meaningful improvement in disease activity: DAS28 reduction of at least 1.2 units, low disease activity (DAS28 </= 3.2) or remission (DAS28 <2.6) | approximately 3 years
Clinical/demographic patient characteristics at initiation of RoActemra/Actemra treatment | approximately 3 years
Treatment regimens: Concomitant medications | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Safat, Kuwait
- Lebanon (4):
  - Beirut
  - Byblos
  - Saida
  - Tripoli
- Doha, Qatar
- Dubai, United Arab Emirates